CLINICAL TRIAL: NCT02174185
Title: A Prospective and Comparative Study of Health-related Quality of Life (HRQoL) in Patients With Conduit Diversion or Orthotopic Neobladder
Brief Title: Compare the Quality of Life Between Patients With Conduit Diversions or Orthotopic Neobladders
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Zhang Xiaoping, Director of Department of Urology, Wuhan Union Hospital, HUST, Huazhong University of Science and Technology
Other Study IDs: 01-18-530605
Record Dates: First submitted 2014-06-22; First posted 2014-06-25 (Estimated); Last update posted 2014-08-04 (Estimated); Status verified 2014-08

CONDITIONS: Bladder Cancer
Keywords: bladder cancer; conduit diversion; orthotopic neobladder; health-related quality of life; validated questionnaire
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- bladder cancer, conduit diversion: new patients with bladder cancer scheduled for radical cystectomy and subsequent conduit diversion
  Interventions: Behavioral: validated health-related quality of life questionnaires
- bladder cancer, orthotopic neobladder: new patients with bladder cancer scheduled for radical cystectomy and subsequent orthotopic neobladder
  Interventions: Behavioral: validated health-related quality of life questionnaires

INTERVENTIONS:
Behavioral: validated health-related quality of life questionnaires — All eligible patients who agree to participate will be asked to fulfill three different validated health-related quality of life questionnaires (EORTC-QLQ-C30/BLM, FACT-BL and BCI) prior to surgery and at 3, 6, 12, 18 months postoperatively.

SUMMARY:
The aim of this study is to compare the health-related quality of life (HRQoL) between patients underwent conduit diversion and orthotopic neobladder after radical cystectomy. The investigators plan to use validated HRQoL questionnaires to learn about how the different urinary diversion operations affect the HRQoL of people living with bladder cancer. The findings from this study may help doctors and patients choosing the proper operation type.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of muscle invasive bladder cancer
* Must be scheduled for radical cystectomy and subsequent conduit diversion or orthotopic neobladder
* Must be able to provide informed consent
* Must be 18 years of age or older
* May have had received intravesical neoadjuvant, adjuvant chemotherapy or immunotherapy

Exclusion Criteria:

* Follow-up data not obtained at Wuhan Union Hospital

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All eligible patients in Wuhan Union Hospital, Huazhong University of Science and Technology.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2014-08; Primary Completion 2018-08 (Estimated); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in HRQoL of bladder cancer patients with different types of urinary diversions | Preoperative baseline and 3, 6, 12, 18 months postoperatively

SECONDARY OUTCOMES:
Score differences between the two groups of patients in the relevant domains from three various validated tools of HRQoL | Preoperative baseline and 3, 6, 12, 18 months postoperatively
  The aim is to compare three various validated tools of HRQoL to study their relative contributions in accounting for variance in prediction of patient HRQoL.
  The three validated tools of HRQoL are EORTC-QLQ-C30/BLM (The European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire/bladder cancer module), FACT-BL (Functional Assessment of Cancer Therapy-Bladder cancer) and BCI (Bladder Cancer Index).
  The two groups are conduit diversion group and orthotopic neobladder group.
Score changes of each patient group during the follow-up | Preoperative baseline and 3, 6, 12, 18 months postoperatively
  Longitudinally learn about the changes of each individual patient HRQoL after urinary diversion and compare the changes of two groups, i.e. conduit diversion group and orthotopic neobladder group.
Objective examination outcomes | Preoperative baseline and 3, 6, 12, 18 months postoperatively
  Supplement the assessment by interviewing the patients with some lab and image examinations, such as renal function tests, liver function tests, urine culture, urine cytology, chest radiography, ultrasound of kidney, ureter and bladder (KUB) etc.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoping Zhang, MD, PhD, Study Director — Department of Urology, Wuhan Union Hospital, Huazhong University of Science and Technology; Hangchuan Shi, MD, Principal Investigator — Department of Urology, Wuhan Union Hospital, Huazhong University of Science and Technology
Locations (1):
- Department of Urology, Wuhan Union Hospital, Huazhong University of Science and Technology, Wuhan, Hubei, China